CLINICAL TRIAL: NCT01553357
Title: A Pilot Study of Lenalidomide and Dexamethasone in Patients With Primary Plasma Cell Leukemia
Brief Title: Lenalidomide and Dexamethasone in Primary Plasma Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Centro di Riferimento Oncologico della Basilicata (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Pellegrino Musto, Onco-Hematology Department Director at IRCCS-CROB Rionero in Vulture, Italy, IRCCS Centro di Riferimento Oncologico della Basilicata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROB0108/1 -- RV-PCL-PI-350; 2008-003246-28 (EudraCT Number)
Record Dates: First submitted 2012-03-03; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Primary Plasma Cell Leukemia
Keywords: Plasma cell leukemia; Lenalidomide; Dexamethasone; Multiple myeloma; Bortezomib; Stem cell transplantation
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide, dexamethasone — Enrolled patients received lenalidomide at a dose of 25 mg/d for 21 days and oral dexamethasone at a dose of 40 mg on days 1, 8, 15, and 22 for each 28-day cycle. After 4 cycles, responding patients not eligible for SCT continued until 8 cycles of full-dose LD, if tolerated, followed by a maintenance dose of single agent lenalidomide equal to 10 mg/d on days 1-21 of each 28-day cycle.
  Patients responding after 4 cycles and eligible for SCT proceeded according to single Centre transplant policy. Patients not responding after 4 cycles or progressing during this treatment were considered off-study.
  Other Names: Revlimid

SUMMARY:
This is an open label, multicenter, exploratory, single arm, two-stage study aiming to explore efficacy and safety of lenalidomide and dexamethasone combination (LD) as first line therapy in previously untreated patients with primary Plasma Cell leukemia (PPCL).

DETAILED DESCRIPTION:
The primary endpoint was response rate according to International Uniform Criteria; secondary endpoints were: i) time to progression (TTP), progression free survival (PFS, and overall survival (OS); ii) percentage of eligible PPCL patients able to mobilize and collect peripheral blood stem cells after LD treatment; iii) percentage of eligible PPCL patients able to undergo autologous or allogeneic stem cells transplantation after LD treatment; iv) serious/severe adverse event (SAEs) rate.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients fulfilling the IMWG diagnostic criteria of PPCL
* Age > 18 years
* ECOG performance status of 0,1 or 2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Myocardial infarction within 6 months prior to enrollment or uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* ECG evidence of acute ischemia or active conduction system abnormalities
* Female subjects either pregnant or breast-feeding
* Serious medical or psychiatric illness
* Total bilirubin greater than 2.0 mg/dL and/or SGOT or SGPT greater than two and a half times normal (unless due to primary malignancy)
* History of severe hepatic dysfunction
* Active infections or HIV positivity
* Uncontrolled insulin-dependent diabetes mellitus
* Uncompensated major thyroid or adrenal dysfunction
* Hemodialysis or peritoneal dialysis
* Renal dysfunction (unless due to primary malignancy; in this case, enrollment at the discretion of the principal investigator)
* ECOG performance status of 3 (unless due to primary malignancy; in this case, enrollment at the discretion of the principal investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 4 months
  IMWG criteria
Complete remission rate | 4 months
  IMWG
At least Very good partial remission rate | 4 months
  IMWG

SECONDARY OUTCOMES:
Progression free survival | 24 months
  Median follow-up
Overall survival | 24 months
  Median follow-up
Percentage of patients able to perform stem cell transplantation | 12 months
  Number of eligible patients reaching stem cell transplantation procedure
Safety | 4-8 months, according to protocol
  Number of severe/serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pellegrino Musto, MD, Principal Investigator — GIMEMA Multiple Myeloma Working Party
Locations (1):
- IRCCS - CROB Ethic Committee, Rionero in Vulture, Pz, Italy